CLINICAL TRIAL: NCT02848820
Title: Initial Non-operative Treatment Strategy Versus Appendectomy Treatment Strategy for Simple Appendicitis in Children Aged 7-17 Years Old - Antibiotics Versus Primary Appendectomy in Children With Simple Appendicitis: APAC Study
Brief Title: Initial Non-operative Treatment Strategy Versus Appendectomy Treatment Strategy for Simple Appendicitis in Children
Acronym: APAC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ramon Gorter (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Amsterdam UMC, location VUmc (Other)
Responsible Party: Sponsor-Investigator, Ramon Gorter, drs., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APAC2016
Record Dates: First submitted 2016-07-24; First posted 2016-07-29 (Estimated); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Appendicitis
Keywords: Appendicitis; Appendectomy; Antibiotics
MeSH Terms: conditions — Appendicitis | interventions — Amoxicillin-Potassium Clavulanate Combination; Gentamicins; Amoxicillin; Clavulanic Acid; Appendectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Augmentin + Gentamicin (Experimental): Initial non-operative treatment strategy reserving an appendectomy for those not responding or with recurrent disease. It consist of:
  Clinical observation for 48 hours with administration of Intravenous administration of amoxicillin/clavulanic acid 25/2.5mg 6-hourly (total 100/10 mg/kg daily; maximum 6000/600mg a day) and gentamicin 7mg/kg once daily for 48 hours. If after 48 hours the patient fulfils the predefined discharge criteria, the antibiotics will be switched to oral amoxicillin/clavulanic acid 50/12.5 mg/kg 8-hourly (max 1500/375mg a day) for in total 7 days and discharge. An appendectomy is reserved for those patients with clinical deterioration, non-improvement after 72 hours or recurrent appendicitis.
  Pain medication according to national protocol.
  Interventions: Drug: Augmentin + Gentamicin
- Operative treatment strategy (Active Comparator): Clinical observation and semi-urgent appendectomy. Pre-, peri- and postoperative care according to local protocol. No routine postoperative antibiotics. Discharge if the patient fulfils the predefined discharge criteria. Pain medication according to national protocol.
  Interventions: Procedure: Appendectomy

INTERVENTIONS:
Drug: Augmentin + Gentamicin — Amoxicillin/clavulanic acid (Augmentin) 25/2.5mg 6-hourly (total 100/10 mg/kg daily; maximum 6000/600mg a day) intravenously for 48 hours Oral amoxicillin/clavulanic acid 50/12.5 mg/kg 8-hourly (max 1500/375mg a day) for in total 7 days Gentamicin 7mg/kg once daily for 48 hours
  Other Names: Amoxicillin/clavulanic acid (Augmentin) + Gentamicin
  Arms: Augmentin + Gentamicin
Procedure: Appendectomy — Pre-, peri- and postoperative care according to local protocol. No routine postoperative antibiotics
  Arms: Operative treatment strategy

SUMMARY:
OBJECTIVE

The aim of this study is to compare the effectiveness of initial non-operative treatment strategy (reserving appendectomy for those not responding or with recurrent disease) with immediate appendectomy in children from 7 to 17 years old, inclusive, with acute simple appendicitis in terms of complications, health-related QOL and costs.

Main research question: What is the difference in proportion of patients experiencing complications within 1 year between both strategies in children from 7 to 17 years old, inclusive, with acute simple appendicitis?

DETAILED DESCRIPTION:
Initial non-operative treatment of acute simple appendicitis has recently been investigated in both the adult as the paediatric population. In the adult population, six Randomised Controlled Trial (RCTs) showed that an appendectomy could be avoided in 40-76% of the patients at the end of their follow-up period. Despite the fact that some patients need to undergo a delayed appendectomy, it has been demonstrated in systematic reviews that non-operative treatment strategy is associated with a significant reduction in complications, faster recovery and return to work, less pain duration and analgesic medication consumption. In children only pilot data is yet available. Short-term success rates of this strategy (including of the investigators own pilot cohort study) are between the 83-92%. Long-term results (one-year follow-up) are available from two studies; 62-75% did not require an appendectomy. No large RCT have yet been conducted in the paediatric population. It is therefore essential to generate high quality empirical evidence regarding this strategy in this subset of patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 7-17 years
* Radiologically confirmed simple appendicitis, defined as:

  1. Clinical findings:

     * Unwell, but not generally ill
     * Localized tenderness in the right iliac fossa region
     * Normal/hyperactive bowel sounds
     * No guarding
     * No mass palpable
  2. Ultrasonography:

     * Incompressible appendix with an outer diameter of ≥6 mm
     * Hyperaemia within the appendiceal wall
     * Without faecolith
     * Infiltration of surrounding fat
     * No signs of perforation
     * No signs of intra-abdominal abscess/phlegmon

Exclusion Criteria:

* Generalized peritonitis, complex appendicitis or sepsis (based upon predefined criteria and scoring system).
* Scoring system: As scoring system was developed determining the risk of complex appendicitis based upon five pre-operative variable. Points have been awarded to each variable. In case the total score is less than 4 points, the patient is likely to have a simple appendicitis. In case the score is 4 or more points, the chance of having complex appendicitis is significant and those children will be excluded from this study. Variables:

  * Diffuse abdominal guarding (3 points)
  * C-Reactive Protein level more than 38 mg/L (2 points)
  * Signs on ultrasound indicative of complex appendicitis (2 points)
  * More than one day abdominal pain (2 points)
  * Temperature: more than 37.5 degree Celsius (1 point)
* Faecolith (ultrasound)
* Serious co-morbidity
* Recurrent appendicitis
* Suspicion of an underlying malignancy or inflammatory bowel disease
* Documented type 1 allergy to the antibiotics used.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 302 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients experiencing complications | One year follow up

SECONDARY OUTCOMES:
Number of days absent from school, social or sport events | 7 days, 1,6,12 months
Number of days absent from work | 7 days, 1,6,12 months
Total number of extra visits (not the already scheduled ones) to the outpatient clinic, general practitioners office or emergency department for abdominal pain. | 7 days, 1,6,12 months
Total length of hospital stay during the follow-up period for strategy related treatment or complications | 7 days, 1,6,12 months
Total days of analgesics medication use. | one month
Pain score measured by the Visual Analogue Scale (VAS) | Clinical phase (up to 7 days)
Proportion of patients with missed diagnosis of complex appendicitis with risk of peritonitis | 7 days, 1,6,12 months
Proportion of patients not having to undergone appendectomy | 7 days, 1,6,12 months
Proportion of patients experiencing recurrent appendicitis | 7 days, 1,6,12 months
Proportion of patients experiencing early failure of initial non-operative treatment. | 7 days, 1,6,12 months
Proportion of patients that undergo interval appendectomy. | 7 days, 1,6,12 months
Quality of life questionnaire (CHQ-CF87, EQ-5d-Youth, EQ-5d-Proxy) | 7 days, 1,6,12 months
Medical and non-medical costs (Health and Labor questionnaire) | 1,6,12 months
Quality adjusted life years (QALY's). Calculating using outcome 13 and 14 | 1,6,12 months
Patient satisfaction questionnaire (PSQ-18 & Net promotor score) | 7 days, 1,6,12 months
Promoting and obstructing factors of implementability measured by questionnaires | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ernst van Heurn, MD PhD, Study Chair — Pediatric Surgical Center of Amsterdam (VUmc & AMC); Ramon Gorter, MD, Study Director — Pediatric Surgical Center of Amsterdam (VUmc & AMC); Roel Bakx, MD PhD, Principal Investigator — Pediatric Surgical Center of Amsterdam (VUmc & AMC)
Locations (15):
- Netherlands (15):
  - Medical Center Alkmaar, Alkmaar
  - Flevoziekenhuis, Almere Stad
  - Amstelland, Amstelveen
  - AMC, Amsterdam
  - OLVG, Amsterdam
  - VU University medical center, Amsterdam
  - Gelre Hospital, Apeldoorn
  - Rijnstate, Arnhem
  - Red Cross Hospital, Beverwijk
  - Albert Schweitzer, Dordrecht
  - Maxima medical center, Eindhoven
  - Zuyderland, Heerlen
  - Antonius Hospital, Nieuwegein
  - Franciscus, Gasthuis en Vlietland, Rotterdam
  - Haga ziekenhuis, The Hague

IPD SHARING:
Plan to Share IPD: Undecided
Will follow

REFERENCES:
- [Derived] Knaapen M, van der Lee JH, Bakx R, The SL, van Heurn EWE, Heij HA, Gorter RR; APAC collaborative study group. Initial non-operative management of uncomplicated appendicitis in children: a protocol for a multicentre randomised controlled trial (APAC trial). BMJ Open. 2017 Nov 15;7(11):e018145. doi: 10.1136/bmjopen-2017-018145. PMID 29146647